CLINICAL TRIAL: NCT00755157
Title: A Phase II Study of the Combination of Metronomic Docetaxel and Bevacizumab as 2nd Line Treatment in Patients With Small Cell Lung Cancer (SCLC)
Brief Title: Metronomic Docetaxel and Bevacizumab in Patients With Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Vassilis Georgoulias, MD, MD, University Hospital of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.06
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Small Cell Lung Cancer
Keywords: Cancer; SCLC; Docetaxel; Bevacizumab; Chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — Docetaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Docetaxel(metronomic)/Bevacizumab
  Interventions: Drug: Docetaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Docetaxel — Metronomic docetaxel (IV) 30 mg/m2 on days 1, 8, 15 every 4 weeks for 6 cycles maximum
  Other Names: Taxotere
Drug: Bevacizumab — Bevacizumab (IV) 10 mgr/Kgr on day 1 and 15 every 4 weeks for 6 cycles maximum followed by (not compulsory) Bevacizumab (IV) 10 mgr/Kgr on day 1 and 15 every 4 weeks until disease progression
  Other Names: Avastin

SUMMARY:
This trial will evaluate the efficacy and safety of metronomic docetaxel and bevacizumab combination in patients with pretreated, advanced small cell lung cancer.

DETAILED DESCRIPTION:
Approximately 80% of the patients with localized SCLC and all of the patients with extensive SCLC will relapse after 1st line chemotherapy. For the chemo-resistant patients (eg those that have relapsed during or less than 3 months after 1st line chemotherapy the sole agent approved for 2nd line chemotherapy is topotecan. Docetaxel has shown some activity as 1st line treatment (ORR 17%). The low dose metronomic chemotherapy that is administered in short intervals has been shown in vitro an in vivo to have antiangiogenic effects. Bevacizumab is a well known anti-angiogenic agent. Recently, a phase III study of 1st line treatment in patients with advanced or metastatic NSCLC showed that the addition of bevacizumab to a platinum-based regimen provided a survival benefit. A number of phase II studies are currently evaluating the addition of bevacizumab to 1st line chemotherapy in SCLC patients with promising results of safety and efficacy. Given the poor results of 2nd line chemotherapy in SCLC we feel that the evaluation of the combination of metronomic docetaxel and bevacizumab (2 anti-angiogenic agents) in such patients is justified. This study will evaluate the combination of metronomic docetaxel and bevacizumab as 2nd line treatment of SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, metastatic (stage IV) small cell lung cancer
* One previous chemotherapy regimen metastatic SCLC
* Measurable disease, defined as at least 1 bidimensionally measurable lesion ≥ 20 X 10 mm
* Age ≥ 18 years
* Performance status (WHO) 0-2
* Life expectancy of at least 12 weeks
* Adequate bone marrow (ANC ≥ 1,500/mm3, PLT ≥ 100,000/mm3, Hgb ≥ 11 g/dL), liver (Bilirubin ≤ 1.5 upper normal limit, SGOT/SGPT ≤ 2.5 upper normal limit in the absence of liver metastases or ≤ 5 upper normal limit in the presence of liver metastases), and renal function (Creatinine ≤ 1,5 upper normal limit)
* Patients must be able to understand the nature of this study and give written informed consent

Exclusion Criteria:

* Second primary malignancy, except for non-melanoma skin cancer
* Pregnant or lactating women
* Any serious, uncontrolled comorbidity on the investigator's judgment
* Uncontrolled infection
* Any sustained chronic toxicity > grade 2 according to the NCI CTCAE (version 3.0)
* Brain metastases, except if radiated and asymptomatic
* Radiotherapy within the previous 4 weeks
* Previous radiotherapy to the only measurable lesion
* Proteinuria ≥ 500 mgr of protein daily
* Hemoptysis > 10 cc per event
* Clinically significant hematemesis
* Centrally located lesion or in contact with major vessels
* Pulmonary lesion with cavitation
* Documented hemorrhagic diathesis or coagulation disorder
* Cardiovascular disease (class II-IV NYHA congestive heart failure, myocardial infarction within the previous 4 months, unstable angina, LVEF < normal, ventricular arrhythmia, uncontrolled hypertension)
* Thrombotic event within the previous 6 months
* Concurrent use of aspirin > 325 mgr daily, low molecular weight heparin in therapeutic dose, warfarin or acenocoumarol, non-steroid anti-inflammatory agents
* Concurrent treatment with other anti-cancer drug
* Major surgical procedure within the previous 4 weeks
* Serum Να+ < 120 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | up to 6 months

SECONDARY OUTCOMES:
Progression free survival | 1 year
Toxicity profile | Toxicity assessment at every cycle
Overall Survival | 1 year
Quality of life assessment | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Agelaki, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (3):
- Greece (3):
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens